CLINICAL TRIAL: NCT03758261
Title: Randomized Clinical Trial of Erector Spinae Plane (ESP) Versus Paravertebral Nerve (PVB) Blockade for Video Assisted Thoracoscopic Surgery (VATS)
Brief Title: Erector Spinae Plane vs. Paravertebral Nerve Block for Thoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Luke (Other)
Responsible Party: Sponsor-Investigator, Charles Luke, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO18070064
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Thoracic Surgical Procedures
Keywords: VATS; Regional Anesthesia; Paravertebral nerve block; Erector Spinae nerve block; Video assisted thoracoscopic surgery

STUDY DESIGN:
Intervention Model Description: 2 groups of patients will be studied simultaneously. One group will have the intervention of the nerve block in the erector spinae approach and the other group will have the nerve block in the traditional paravertebral approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Nerve Block (Other): Erector Spinae nerve block
  Interventions: Drug: Erector Spinae nerve block
- Paravertebral Nerve Block (Other): Paravertebral nerve block
  Interventions: Drug: Paravertebral nerve block

INTERVENTIONS:
Drug: Paravertebral nerve block — The patient will be placed in a sitting position and the level of needle insertion will be marked corresponding to the level of surgical incision. With sterile technique an ultrasound Paravertebral Nerve Block will be performed.
  Arms: Paravertebral Nerve Block
Drug: Erector Spinae nerve block — The patient will be placed in a sitting position and the level of needle insertion will be marked corresponding to the level of surgical incision. With sterile technique an ultrasound erector spinae nerve block will be performed.
  Arms: Erector Spinae Nerve Block

SUMMARY:
Continuous paravertebral analgesia and erector spinae plane blockade (ESP) are accepted techniques at University of Pittsburgh Medical Center (UPMC) for the management of thoracic pain following surgery and trauma. Recently, an increasing number of erector spinae plane nerve blocks are being performed as it has been demonstrated in our institution, and via case reports that the blocks provide clinical effectiveness, but may have a better side-effect profile than the paravertebral nerve block. However, the relative efficacy of ESP compared to paravertebral nerve block remains to be established for video assisted thoracoscopic surgery (VATS). This is a prospective randomized study intended to assess the efficacy, safety and side-effect profile of continuous erector spinae plane analgesia versus continuous paravertebral analgesia for VATS procedures. It will include 60 patients presenting to UPMC Passavant for a VATS procedure. Patients will be randomized 1:1 to receive either a nerve block via continuous paravertebral infusion or via erector spinae plane infusion. In addition, to treat breakthrough pain, the patients in both arms will receive multimodal adjunctive therapy per routine. Bupivacaine and ropivacaine are FDA approved for use in nerve block catheters. The primary outcome will be to compare analgesic efficacy between the two nerve blocks as defined by total opioid consumption and pain scores on the numeric pain rating scale. Secondary outcomes include incentive spirometer amounts (baseline vs daily score postoperatively), length of stay, duration of catheter and report of adverse events or complications. Other data points include number of chest tubes and location and level of catheter and nerve block placement as well as number of blocks per case.

DETAILED DESCRIPTION:
Background and significance:

Multimodal analgesia for thoracic surgery is key to allow faster recovery and diminish postoperative complications. Paravertebral nerve blocks as well as epidurals are among the regional anesthetic techniques utilized for these procedures. Recently, a newer technique, the erector spinae plane block, has been used and described to be effective in treating pain for patients undergoing thoracic surgery. At UPMC, the investigators have had clinically significant pain control for thoracic surgery with both types of blocks. The previous case reports/series and our clinical observation has led us to propose this study of comparing the clinical efficacy of erector spinae plane block vs. paravertebral nerve block.

Though ESP and paravertebral blocks have been documented to be efficacious for this procedure, there has been no direct comparison between the two approaches. The ESP block is considered to be a safer technique with less theoretical adverse events possible and thus, would become a viable alternative to the more technically challenging paravertebral nerve block. If ESP is found to be superior or non-inferior to paravertebral in terms of pain management and safety, this would be a major finding, as ESP is considered safer and technically easier to perform than paravertebral nerve block.

Study design and methods

The investigators present a prospective randomized trial comparing the efficacy of continuous paravertebral nerve blocks vs. ESP blocks for video assisted thoracoscopy surgery (VATS) at UPMC Passavant.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing VATS agreeable to have a nerve block as analgesic technique
* Age: 18 years old and older.
* ASA (American Society of Anesthesiologists Class) I-IV

Exclusion criteria:

* Cognitive impairment that would not allow effective nerve block placement or gathering information related to the study (ex. pain score).
* Contraindications for nerve block placement such as coagulopathy, use of clopidogrel in the past 48hs, patients on dual antiplatelet therapy, infection at the site of puncture, patient refusal, allergy to local anesthetics.
* Chronic opiate consumption
* Patient expected to be on therapeutic anticoagulation post procedure.
* Pregnancy
* Comorbid conditions: Any comorbid condition that in the judgment of the anesthesiologist would preclude the patient from any aspect of the study (ex. sepsis, possibly abnormalities of the thoracic spine or paravertebral anatomy such as neoplastic mass occupying the space, empyema, increased intracranial pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Luke, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Passavant, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experiences of ultrasound-guided erector spinae plane block for thoracic vertebra surgery. J Clin Anesth. 2017 May;38:137. doi: 10.1016/j.jclinane.2016.12.028. Epub 2017 Feb 17. No abstract available. PMID 28372654 (Retraction: PMID 35396111 J Clin Anesth. 2022 Aug;79:110791)
- [Background] Luis-Navarro JC, Seda-Guzman M, Luis-Moreno C, Lopez-Romero JL. The erector spinae plane block in 4 cases of video-assisted thoracic surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Apr;65(4):204-208. doi: 10.1016/j.redar.2017.12.004. Epub 2018 Jan 11. English, Spanish. PMID 29336785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Started | 17 | 16
Completed | 15 | 15
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.47 (13.51) | 65.94 (12.22) | 65.18 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33
Weight (kg) [Mean (Standard Deviation); unit: kilogram (kg)] | 79.98 (23.04) | 80.17 (17.79) | 80.07 (20.66)
Height (cm) [Mean (Standard Deviation); unit: centimeter (cm)] | 167.35 (9.90) | 165.21 (8.69) | 166.31 (9.39)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.54 (8.33) | 29.49 (5.96) | 29.00 (7.29)

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption
Description: Morphine equivalents (total OME)
Time Frame: 1 day post catheter removal
Measure: Mean (Standard Deviation); unit: mg morphine equivalent (MME)
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
mg morphine equivalent (MME) | 187.36 (184.35) | 164.70 (142.64)

2. Primary Outcome: Patient Reported Pain Scores
Description: Visual analog scale. Scale is from 0 to 10 numerical pain rating scale. 0 indicates no pain. 10 indicates maximum level of pain. Higher scores indicate worse pain level. Pain score will be a single number from 0 to 10.
Time Frame: 1 day post catheter removal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
score on a scale | 5.98 (2.21) | 5.16 (2.66)

3. Secondary Outcome: Amount Achieved on Incentive Spirometer
Description: Amount achieved on incentive spirometer device (mL). Higher level indicates better respiratory effort
Time Frame: 1 day post catheter removal
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
milliliter (mL) | 1221.15 (480.77) | 1187.50 (541.27)

4. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay post-surgery
Time Frame: Up to 2 weeks on average
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
hours | 101.96 (49.99) | 96.30 (41.78)

5. Secondary Outcome: Time Catheter Remains Inserted in Body
Description: How long catheter remains providing pain relief
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
hours | 21.99 (12.96) | 21.94 (11.91)

6. Secondary Outcome: Averaged Total of Narcotic Usage
Description: Averaged total Narcotic consumption measured in Oral Morphine Equivalence (OME)
Time Frame: 0-120 hours post-operative
Measure: Mean (Standard Deviation); unit: Average of OME
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
Average of OME | 187.36 (190.82) | 164.7 (147.64)

7. Secondary Outcome: Report of Adverse Events From Catheter Placement
Description: Participant count for patients who experienced adverse events with nerve block catheter placement which includes pneumothorax, infections, bleeding, local anesthetic toxicity.
Time Frame: 1 day post catheter removal
Measure: Count of Participants; unit: Participants
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of admission until patient discharge, an average of 4-days.
Arm/Group | Erector Spinae Nerve Block | Paravertebral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erector Spinae Nerve Block (N=17) | Paravertebral Nerve Block (N=16)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Respiratory Depression
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) — Patient went into atrial fibrillation.
Redo Nerve Block (Surgical and medical procedures) | 0 (0) | 1 (1) — The patient's nerve block had to be redone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT03758261/Prot_003.pdf
  • Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT03758261/SAP_004.pdf
  • Informed Consent Form (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT03758261/ICF_002.pdf